CLINICAL TRIAL: NCT03103139
Title: Randomized Controlled Trial Of Endoscopic Stenting Across the Papilla Versus the Leak Site to Treat Bile Leak
Brief Title: Endoscopic Stenting Across the Papilla Versus the Leak Site to Treat Bile Leak
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, James Buxbaum, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-16-00520
Record Dates: First submitted 2016-12-07; First posted 2017-04-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Bile Leak

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transpapillary Stents (Active Comparator): Stent placement across the Papilla (with a short plastic stent) for biliary leak
  Interventions: Procedure: Transpapillary Stent
- Stent across bile leak (Experimental): Stent placement across the bile leak (with a longer stent) for biliary leak
  Interventions: Procedure: Stent across bile leak

INTERVENTIONS:
Procedure: Transpapillary Stent — ERCP with placement of short stent
  Arms: Transpapillary Stents
Procedure: Stent across bile leak — ERCP with long stent
  Arms: Stent across bile leak

SUMMARY:
1. Biliary duct injury are a relatively frequent complication of hepatobiliary surgery, most comonly laparoscopic cholecystecomy.
2. Prior to the development of more sophisticated endoscopic interventions, repeat surgery was often necessary for the management of biliary leaks.
3. Advances in technique and technology in gastroenterology endoscopy have largely replaced surgery as the first line intervention for biliary leak.
4. Most practices utilize endoscopic plastic biliary stent placement alone and are efficacious and equivalent to the biliary stent placement with endoscopic biliary sphincterotomy.
5. An area of variation is in whether biliary stent should cross the papilla ( with a shorter stent) versus the site of the bile leak (with a longer stent).
6. Our objective is to assess whether placing a biliary stent across the leak versus across the papilla alone improves the treatment of biliary leaks.

DETAILED DESCRIPTION:
1.0 BACKGROUND 1.1) Biliary duct injuries are a relatively frequent complications of hepatobiliary surgery, most commonly laparoscopic cholecystectomy1. Such injuries can manifest clinically in a number of ways including biliary leakage, biliary stricture formation, or associated infectious complications. Biliary leakage is the most common of these postoperative complications and is estimated to be clinically significant in 0.8 to 1.1% of such surgeries.

Prior to the development of more sophisticated endoscopic interventions, repeat surgery was often necessary for management of biliary leaks. However, advances in technique and technology in gastrointestinal endoscopy have largely replaced surgery as a first line intervention for biliary leaks. The generally accepted goal in the endoscopic management of biliary leaks is to equalize the pressure between the biliary system and the duodenum, so as to allow bile to flow into the lower pressure small bowel and thereby affording the leak time to close.

How to best achieve this goal has been a topic of considerable interest. Randomized studies have shown that endoscopic plastic biliary stent placement alone is highly efficacious and equivalent to biliary stent placement with endoscopic biliary sphincterotomy. Thin (7 French[Fr]) and wide (10 French) diameter stents seem to have similar efficacy with regards to leak resolution. Beyond these well-validated techniques, there are other variations in clinical practice that are not supported by high-levels of evidence.

1.2) One area of variation is in whether the biliary stent should cross the papilla (with a shorter stent) versus the site of the leak (with a longer stent).

2.0 OBJECTIVES AND PURPOSE

To assess whether placing a biliary stent across the leak versus across the papilla alone improves the treatment of biliary leaks.

3.0 STUDY DESIGN:

The study will be a prospective randomized controlled trial. All patients undergoing Endoscopic Retrograde Cholangiopancreatography (ERCP) for the treatment of bile leaks will be eligible for inclusion (see section and initial collection form). During the ERCP if cholangiogram demonstrates a leak, the patient will be randomized to either A) papillary stenting strategy or B) crossing the leak site strategy. Please see the diagram below to complement the written description of the study design.

A) In the papillary stenting strategy, regardless of where the leak is identified, a stent is placed into the duodenal papilla and into the most distal (proximal to duodenum) portion of the bile duct. The goal of this strategy is to use the stent to keep the papilla open, thereby decreasing the pressure gradient and allowing for bile to flow preferentially into the duodenum away from the leaking area. All stents in this strategy will be 7 Fr in diameter and 5 cm long.

B) In the crossing the leak strategy (left), once the area of bile leakage is identified in the biliary tree, a stent will be placed endoscopically across the leaking area. This theoretically allows the underlying injured bile duct tissue to heal. The same diameter stent (7Fr) as the papillary stenting strategy will be used but the length will vary in order to bridge the leaking region (5-15cm).

The decision whether or not to perform sphincterotomy will be entirely determined by the attending endoscopist and not part of the study. The 7Fr stents we are using may be easily placed whether or not a sphincterotomy is performed. It will be recorded whether or not a sphincterotomy was performed. All procedures evaluated in this study are done as part of standard clinical care.

Following the initial ERCP intervention, the patients will receive routine post-procedural care. They will have serial monitoring.

CRITERIA FOR EVALUATION AND ENDPOINT DEFINITIONS

The primary outcome will be a successful resolution of bile leak with the ERCP strategy. This will require will require 2 criterion:

A. No further leakage of bile on the follow up ERCP at 5 weeks. Resolution is confirmed by the demonstration of no leaking of contrast from the prior leakage site on cholangiography.

B. No ERCP or other procedure has to be done between the initial ERCP and the 5 week ERCP to treat the bile leak.

The proportion of patients in each randomized arm with the resolution of bile leak at 5 weeks will be compared.

.

There will be several secondary outcomes:

A. Time from ERCP to removal of surgical drain (days) B. Time from ERCP to complete cessation of output from drain (days) C. Presence of other significant findings on the 5th week cholangiogram. These include bile duct stone or biliary stricture.

D. Requirement of surgery to treat the bile leak. E. Endoscopic complications of the 1st and 2nd ERCP including pancreatitis, bleeding perforation, cholangitis, and stent occlusion within 5 weeks of initial or 2nd ERCP.

STATISTICAL CONSIDERATONS:

Patients will be randomized in a 1:1 fashion to either the papillary stenting strategy group or crossing the leak stenting strategy group.

Dichotomous outcomes including primary outcome (successful resolution of the bile leakage) will be compared using a Fischer's exact or chi squared test. Continuous baseline charactersistics or outcomes will be compared using a Wilcoxan rank sum test or T test depending on distribution. If imbalances occur, logistic regression models will be developed to control for these imbalances as covariates in the primary outcome model. Secondary outcomes involving time to clinical improvement in the arms will be compared using Cox Regression analysis, allowing for the inclusion of covariates depending on degree of balance of baseline characteristics. Analyses will be performed using SPSS v.23 and SAS v9; two-sided p = 0.05 will be used for primary and secondary outcomes.

Based on a retrospective query of the 32 consecutive previous cases of bile leaks managed at the Los Angeles County hospital using stents which did or did not bridge the leak we used G*Power to estimate that a total sample size of 88 will be adequate (2 sided alpha of 0.05 and beta of 0.2) to detect an 20% difference (80 vs 99%) in successful resolution of bile leak in the two groups. Based on data from the past 1 year at Los Angles County hospital it was estimated that there would be a 5% 5-week attrition thus the sample size was determined to be 92 patients.

DSM (includes biostatistician, independent senior investigator) will review for safety differences and study progress following randomization of 30 and 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ERCP for the treatment of suspected acute bile leaks will be eligible for inclusion (bile leaks felt to be complications of surgical intervention). A patient is suspected to have an acute bile leak if the patient is referred within two weeks following the original surgery.. Legally authorized representatives may serve as surrogates to consent for inclusion in this study.

Bile leaks are suspected based on the following:

A) Persistent, significant drainage of bilious fluid from post-surgical drains following hepatobiliary surgery or cholecystectomy,.

B) Compatible symptoms plus imaging findings on abdominal ultrasonography, computed tomography, HIDA scanning, or MRCP of an abnormal intra-abdominal fluid collection in the setting of recent hepatobiliary surgery.

Exclusion Criteria:

* Patients with bile duct transection (in which the duct has been totally severed into 2 parts) will be excluded as these are known to not be amenable to endoscopic therapy. Further, suspected bile leaks of non-surgical etiology will be excluded from the study (malignancy, trauma, spontaneous perforation, and other rarer causes). Bile leaks suspected two weeks post surgery will also not be included. Additionally patients who are pregnant, imprisoned, under age 18, unable to give informed consent, or have undergone prior biliary diversion surgery will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2016-11; Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with resolution of bile leak by cholangiography | within 5 weeks
  The primary outcome is the proportion of patients with resolution of bile leak determined by cholangiography at 5 weeks among the two groups.

SECONDARY OUTCOMES:
Time to from ERCP to remove surgical drain | within 5 weeks
  The time from the ERCP to removal of surgical drain will be compared in the two groups.
Proportion of patients who required surgery | within 10 weeks
  The proportion of patients who require surgery the manage the bile leaks in the two groups were compared.

CONTACTS AND LOCATIONS:
Overall Officials: James Buxbaum, M.D., Principal Investigator — USC Health Sciences Center
Locations (1):
- Los Angeles County Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buanes T, Waage A, Mjaland O, Solheim K. Bile leak after cholecystectomy significance and treatment: results from the National Norwegian Cholecystectomy Registry. Int Surg. 1996 Jul-Sep;81(3):276-9. PMID 9028989
- [Result] Rossi RL, Schirmer WJ, Braasch JW, Sanders LB, Munson JL. Laparoscopic bile duct injuries. Risk factors, recognition, and repair. Arch Surg. 1992 May;127(5):596-601; discussion 601-2. doi: 10.1001/archsurg.1992.01420050124016. PMID 1533509
- [Result] Barkun AN, Rezieg M, Mehta SN, Pavone E, Landry S, Barkun JS, Fried GM, Bret P, Cohen A. Postcholecystectomy biliary leaks in the laparoscopic era: risk factors, presentation, and management. McGill Gallstone Treatment Group. Gastrointest Endosc. 1997 Mar;45(3):277-82. doi: 10.1016/s0016-5107(97)70270-0. PMID 9087834
- [Result] Davids PH, Ringers J, Rauws EA, de Wit LT, Huibregtse K, van der Heyde MN, Tytgat GN. Bile duct injury after laparoscopic cholecystectomy: the value of endoscopic retrograde cholangiopancreatography. Gut. 1993 Sep;34(9):1250-4. doi: 10.1136/gut.34.9.1250. PMID 8406163
- [Result] Fasoulas K, Zavos C, Chatzimavroudis G, Trakateli C, Vasiliadis T, Ioannidis A, Kountouras J, Katsinelos P. Eleven-year experience on the endoscopic treatment of post-cholecystectomy bile leaks. Ann Gastroenterol. 2011;24(3):200-205. PMID 24713781
- [Result] Bjorkman DJ, Carr-Locke DL, Lichtenstein DR, Ferrari AP, Slivka A, Van Dam J, Brooks DC. Postsurgical bile leaks: endoscopic obliteration of the transpapillary pressure gradient is enough. Am J Gastroenterol. 1995 Dec;90(12):2128-33. PMID 8540501
- [Result] Mavrogiannis C, Liatsos C, Papanikolaou IS, Karagiannis S, Galanis P, Romanos A. Biliary stenting alone versus biliary stenting plus sphincterotomy for the treatment of post-laparoscopic cholecystectomy biliary leaks: a prospective randomized study. Eur J Gastroenterol Hepatol. 2006 Apr;18(4):405-9. doi: 10.1097/00042737-200604000-00014. PMID 16538112
- [Result] Katsinelos P, Kountouras J, Paroutoglou G, Chatzimavroudis G, Germanidis G, Zavos C, Pilpilidis I, Paikos D, Papaziogas B. A comparative study of 10-Fr vs. 7-Fr straight plastic stents in the treatment of postcholecystectomy bile leak. Surg Endosc. 2008 Jan;22(1):101-6. doi: 10.1007/s00464-007-9381-y. Epub 2007 May 22. PMID 17516115
- [Result] Nawaz H, Papachristou GI. Endoscopic treatment for post-cholecystectomy bile leaks: update and recent advances. Ann Gastroenterol. 2011;24(3):161-163. No abstract available. PMID 24713786